CLINICAL TRIAL: NCT00218192
Title: A Trial to Reduce Hepatitis C Among Injection Drug Users
Brief Title: A Trial to Reduce Hepatitis C Among Injection Drug Users - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Stein, MD, PI, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-13759-1; R01DA013759 (NIH); R01-13759-1
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2013-04

CONDITIONS: HCV Negative Status; HCV Risk Behavior
Keywords: hepatitis c; injection drug use
MeSH Terms: conditions — Hepatitis C | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to examine the efficacy of a brief motivational intervention on the cumulative incidence of Hepatitis C.

DETAILED DESCRIPTION:
Injection drug users are at high risk for blood-borne viral infections during their first years of injecting when they are least likely to seek formal substance abuse treatment, and are likely to be practicing risky drug-use behaviors. Research has demonstrated that a brief motivational intervention that includes booster sessions and addresses drug and sex risks is effective in reducing HIV risk behaviors among injection drug users.

Because Hepatitis C Virus is a bloodborne pathogen like HIV, and transmission occurs via similar behaviors, successful HIV prevention strategies should be robust in preventing HCV but need to be tested. Motivational interventions, which aim to elicit a goal and plan from the patient to reduce injection and sexual risk taking, are particularly suited to address behaviorally-based changes. Motivational interventions are individualized and tailored to the risks and concerns of the participant, but can be standardized and evaluated to make this technique applicable in a variety of settings. The occurrence of injection drug use in a population with traditionally poor linkage to primary care, an enormous burden of illness, and high HCV and other blood-borne pathogen transmission risk, supports the use of motivational interventions in this group.

Comparison(s): Participants are assigned, in this 24 month longitudinal study, to an assessment-only condition or an assessment plus motivational intervention condition. Participants in the intervention condition receive up to 4 sessions of motivational interviewing during the first 6 months of the study.

ELIGIBILITY:
Inclusion Criteria:

* current opiate or cocaine use
* HCV seronegative
* able to complete the study procedures in English

Exclusion Criteria:

* current enrollment in a formal substance abuse treatment program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2000-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Hepatitis C seroconversion

SECONDARY OUTCOMES:
Substance use

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, M.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Stein MD, Herman DS, Anderson BJ. A trial to reduce hepatitis C seroincidence in drug users. J Addict Dis. 2009 Oct;28(4):389-98. doi: 10.1080/10550880903183034. PMID 20155608